CLINICAL TRIAL: NCT01835015
Title: A Multi-Center, Open-Label, Single Ascending Dose Study To Assess the Safety, Tolerability, and Serum Pharmacokinetics of Intravitreal CLG561 in Subjects With Advanced Age-Related Macular Degeneration
Brief Title: Pharmacokinetics of CLG561 in Patients With Advanced Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C-12-074
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Age-related Macular Degeneration
Keywords: First in human; Safety; Tolerability; Serum PK; Intravitreal (IVT); Age-related macular degeneration; AMD; Geographic Atrophy; Choroidal neovascularization
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy; Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CLG561, Concentration Level A (Experimental): Single 50 μL intravitreal injection of CLG561, Dose Level A
  Interventions: Drug: CLG561
- CLG561, Concentration Level B (Experimental): Single 50 μL intravitreal injection of CLG561, Dose Level B
  Interventions: Drug: CLG561
- CLG561, Concentration Level C (Experimental): Single 50 μL intravitreal injection of CLG561, Dose Level C
  Interventions: Drug: CLG561
- CLG561, Concentration Level D (Experimental): Single 50 μL intravitreal injection of CLG561, Dose Level D
  Interventions: Drug: CLG561
- CLG561, Concentration Level E (Experimental): Single 100 μL intravitreal injection of CLG561, Dose Level E
  Interventions: Drug: CLG561

INTERVENTIONS:
Drug: CLG561 — Administered by intravitreal injection, Day 1

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and serum pharmacokinetics of CLG561 in subjects with advanced age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Subjects were divided into 5 cohorts, with the subjects in each cohort being administered a single IVT dose of CLG561 in 1 of 5 concentration levels A-E, where A=lowest and E=highest. All subjects received active CLG561. Progress from one cohort to the next was time-lagged to allow for safety review. Dosing was also time-lagged within each cohort. Only one eye (designated as the study eye) was dosed per subject. Post-dose safety assessments and ocular examination occurred immediately after the IVT injection and continued throughout the outpatient visits at pre-determined timepoints. Collection of post-injection blood samples began after the IVT injection at pre-determined timepoints. Subjects were followed for up to 84 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related macular degeneration in study eye, as specified in protocol.
* Poor visual acuity in study eye, as specified in protocol.
* Willing to receive meningitis and pneumonia vaccinations at least 2 weeks prior to study treatment.
* Females must be post-menopausal and/or surgically sterile.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Treatments to the study eye within 28 days prior to study treatment, as specified in protocol.
* Any disease or medication expected to cause systemic or ocular immunosuppression.
* Participation in another interventional clinical study or use of any experimental treatment for AMD within 12 weeks prior to study treatment.
* Other protocol-defined exclusion criteria may apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Sciences, CA CSI NS/Opth, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 investigational centers located in the US.
Pre-assignment Details: Of the 50 enrolled,19 subjects were exited as screen failures prior to randomization. This reporting group includes all assigned subjects (31).
Groups:
- CLG561, Level A: Single 50 μL intravitreal injection of CLG561, Dose Level A
- CLG561, Level B: Single 50 μL intravitreal injection of CLG561, Dose Level B
- CLG561, Level C: Single 50 μL intravitreal injection of CLG561, Dose Level C
- CLG561, Level D: Single 50 μL intravitreal injection of CLG561, Dose Level D
- CLG561, Level E: Single 100 μL intravitreal injection of CLG561, Dose Level E
Period: Overall Study
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Started | 6 | 6 | 7 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled subjects who received CLG561.
Groups:
- Total: Total of all reporting groups
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (6.82) | 76.2 (8.80) | 76.1 (6.69) | 73.3 (9.52) | 76.5 (10.86) | 75.3 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 4 | 5 | 3 | 19
  Male | 0 | 5 | 3 | 1 | 3 | 12
Primary Diagnosis [Number; unit: participants] — Geographic atrophy was classified as atrophic lesions in the macula related to AMD as assessed by Fundus autofluorescence. Exudative (wet) macular degeneration was classified as patients suffering from neovascular (wet) AMD, as assessed by fluorescein angiography, who were not likely to require anti-VEGF (vascular endothelial growth factor) therapy during the study period.
  participants
    Geographic atrophy | 0 | 2 | 2 | 1 | 2 | 7
    Exudative macular degeneration | 6 | 4 | 5 | 5 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) by Visit - Study Eye
Description: BCVA (with spectacles or other visual corrective devices) using Early Treatment Diabetic Retinopathy Study (ETDRS) testing was reported in letters read correctly. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 2, Day 4, Day 15, Day 29, Day 57, Day 85
Population: This analysis population includes all enrolled subjects who received investigational product. Here, "n" is the number of subjects with non-missing values at the specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
letters
  Baseline, n=6,6,7,6,6 | 23.7 (16.55) | 25.7 (15.20) | 27.6 (17.67) | 41.5 (20.42) | 38.0 (11.75)
  Change from Baseline, Day 2, n=6,6,7,6,6 | 0.7 (8.24) | 2.5 (5.24) | 1.1 (3.02) | 0.0 (5.73) | -1.0 (10.02)
  Change from Baseline, Day 4, n=6,6,7,6,6 | 3.5 (8.53) | 4.8 (4.67) | 1.7 (3.04) | 1.8 (5.19) | 3.3 (7.87)
  Change from Baseline, Day 15, n=6,6,6,6,6 | 2.7 (7.99) | 3.7 (4.50) | 2.0 (4.73) | 3.5 (8.26) | 5.2 (8.06)
  Change from Baseline, Day 29, n=6,5,6,6,6 | 2.2 (5.85) | 4.8 (5.02) | 1.3 (5.28) | 2.0 (6.84) | 1.5 (4.51)
  Change from Baseline, Day 57, n=6,5,6,6,6 | 4.7 (11.09) | 2.0 (3.24) | 2.5 (5.75) | 4.2 (11.09) | 2.3 (2.94)
  Change from Baseline, Day 85, n=6,6,6,6,6 | 3.8 (9.43) | 3.0 (4.86) | 2.2 (5.12) | 2.2 (5.12) | 3.2 (5.12)

2. Primary Outcome: Mean Intra-Ocular Pressure (IOP) by Visit - Study Eye
Description: IOP was measured by Goldmann applanation tonometry or tonopen, at the discretion of the Investigator, and reported in mmHg (millimeters of mercury). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 1, Day 2, Day 4, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
mmHg
  Baseline, n=6,6,7,6,6 | 14.7 (2.16) | 14.3 (2.42) | 15.7 (3.86) | 15.2 (3.06) | 16.5 (3.67)
  Day 1, n=6,6,7,6,6 | 16.3 (3.72) | 20.2 (8.01) | 16.6 (6.24) | 22.3 (3.50) | 20.2 (3.97)
  Day 2, n=6,6,7,6,6 | 16.0 (1.79) | 14.5 (1.05) | 14.3 (3.15) | 14.0 (4.00) | 15.0 (3.10)
  Day 4, n=6,6,7,6,6 | 16.2 (2.32) | 14.5 (3.99) | 15.1 (4.74) | 14.7 (4.23) | 15.3 (3.93)
  Day 15, n=6,6,6,6,6 | 14.0 (1.67) | 15.5 (2.81) | 16.2 (6.21) | 16.2 (3.76) | 16.5 (4.09)
  Day 29, n=6,5,6,6,6 | 16.8 (3.19) | 16.8 (4.60) | 16.0 (4.94) | 16.8 (4.26) | 16.2 (4.67)
  Day 57, n=6,5,6,6,6 | 17.7 (2.94) | 15.6 (5.32) | 16.3 (3.27) | 16.3 (2.25) | 15.8 (3.13)
  Day 85, n=6,6,6,6,6 | 16.5 (2.07) | 15.5 (5.24) | 16.7 (4.27) | 16.2 (4.07) | 16.2 (4.26)

3. Primary Outcome: Number of Subjects With Change From Normal to Abnormal in Fundus Examination at Any Post-Therapy Visit as Compared to Baseline Assessment
Description: A dilated fundus examination was performed to evaluate the health of the retina, macula, choroid, and optic nerve. Subjects having a normal baseline evaluation were examined at subsequent visits, and any change from normal to abnormal was recorded. Criteria for reclassifying from normal to abnormal were left to the opinion of the investigators. One eye (study eye) contributed to the analysis. None of the abnormalities were deemed related to the study medication.
Time Frame: Baseline, Day 2, Day 4, Day 8, Day 15, Day 29, Day 57, Day 85
Population: This analysis population includes all enrolled subjects who received investigational product.
Measure: Number; unit: participants
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
participants
  Retina: Baseline Normal | 5 | 4 | 4 | 6 | 5
  Retina: Change from Normal to Abnormal | 1 | 0 | 0 | 0 | 1
  Macula: Baseline Normal | 6 | 6 | 6 | 6 | 6
  Macula: Change from Normal to Abnormal | 0 | 0 | 0 | 0 | 1
  Choroid: Baseline Normal | 6 | 6 | 6 | 6 | 6
  Choroid: Change from Normal to Abnormal | 0 | 0 | 0 | 0 | 0
  Optic Nerve: Baseline Normal | 6 | 3 | 5 | 6 | 5
  Optic Nerve: Change from Normal to Abnormal | 1 | 0 | 2 | 0 | 0

4. Primary Outcome: Number of Subjects With a Change From Normal to Abnormal in Ocular Signs at Any Post-Therapy Visit as Compared to Baseline Assessment
Description: A slit-lamp biomicroscopy examination was performed to evaluate the anterior segment of the eye. Subjects having a normal baseline evaluation were examined at subsequent visits, and any change from normal to abnormal was recorded. Criteria for reclassifying from normal to abnormal were left to the opinion of the investigators. One eye (study eye) contributed to the analysis. None of the abnormalities were deemed related to the study medication.
Time Frame: Baseline, Day 2, Day 4, Day 8, Day 15, Day 29, Day 57, Day 85
Population: This analysis population includes all enrolled subjects who received investigational product.
Measure: Number; unit: participants
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 6
participants
  Lids/Lashes: Baseline Normal | 5 | 4 | 5 | 6 | 6
  Lids/Lashes: Change from Normal to Abnormal | 0 | 1 | 1 | 0 | 1
  Conjunctiva: Baseline Normal | 5 | 4 | 6 | 5 | 5
  Conjunctiva: Change from Normal to Abnormal | 2 | 1 | 4 | 0 | 2
  Cornea: Baseline Normal | 6 | 5 | 6 | 6 | 5
  Cornea: Change from Normal to Abnormal | 0 | 0 | 2 | 0 | 1
  Iris: Baseline Normal | 6 | 6 | 6 | 6 | 6
  Iris: Change from Normal to Abnormal | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Area Under the Serum Concentration-time Curve (AUC) From Time Zero to All [AUC(0-all)]
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method. These data were analyzed using a noncompartmental pharmacokinetic (PK) method.
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: This analysis population includes all subjects who received investigational product, completed at least 1 post-injection study visit and for whom serum concentration-time data is available, provided no collection or analytical deviations which would affect the integrity of the data occurred.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*ng/mL | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | 238000 (81800) | 373000 (160000)

6. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-last)]
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method. These data were analyzed using a noncompartmental PK method.
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*ng/mL | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | 195000 (78300) | 304000 (148000)

7. Secondary Outcome: Time to Reach the Maximum Serum Concentration After Drug Administration (Tmax)
Description: as for outcome 6
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | 144 (62.7) | 187 (79.8)

8. Secondary Outcome: Dose Normalized Observed Maximum Serum Concentration Following Drug Administration (Cmax/D)
Description: as for outcome 6
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL/mg | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | 102 (30) | 75.8 (30.9)

9. Secondary Outcome: Dose-normalized Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-last)/D]
Description: as for outcome 6
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL/mg
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*ng/mL/mg | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | NA (NA) — Statistical analysis was not conducted because the concentration was too low to allow reliable estimation. | 38900 (15700) | 30400 (14800)

10. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Time "t" Where t is a Defined Time Point After Administration [AUC(0-t)]
Description: Serum concentrations at each collection time point were quantitated, where possible, using a validated immunoassay method.
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: This parameter was not calculated as AUClast and AUCall were considered sufficient to characterize the systemic exposure to CLG561.
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Terminal Elimination Half-life (T½)
Description: as for outcome 10
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 10
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: The Apparent Volume of Distribution During the Terminal Elimination Phase Following Extravascular Administration (Vz/F)
Description: as for outcome 10
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 10
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Apparent Systemic (or Total Body) Clearance From Serum Following Extravascular Administration (CL/F)
Description: as for outcome 10
Time Frame: Day 1 pre-injection, 2h, 6h, Day 2, Day 4, Day 6, Day 8, Day 11, Day 15, Day 29, Day 57, Day 85
Population: as for outcome 10
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 84 days). Ocular AEs are presented for both study eye and non-study eye. AEs were obtained as solicited comments and observations by the Investigator.
Description: An AE was defined as any untoward medical occurrence in a subject exposed to study drug or any unfavorable and unintended sign, symptom, or disease temporally associated with use of study drug, or untoward medical occurrence at any time prior to administration of first dose of study drug. AEs were reported as pre-treatment and treatment-emergent.
Groups:
- CLG561, Level A; CLG561, Level B; CLG561, Level C; CLG561, Level D; CLG561, Level E: Reported subsequent to the initiation of treatment
- Pretreatment: Reported prior to the initiation of study treatment
Arm/Group | CLG561, Level A | CLG561, Level B | CLG561, Level C | CLG561, Level D | CLG561, Level E | Pretreatment
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/7 | 0/6 | 0/6 | 0/50
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 6/7 | 2/6 | 3/6 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLG561, Level A (N=6) | CLG561, Level B (N=6) | CLG561, Level C (N=7) | CLG561, Level D (N=6) | CLG561, Level E (N=6) | Pretreatment (N=50)
Blindness Transient (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 — Study Eye.Transient blindness was due to transient rise in intraocular pressure. Visual acuity returned to pre-injection levels after a paracentesis was performed.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLG561, Level A (N=6) | CLG561, Level B (N=6) | CLG561, Level C (N=7) | CLG561, Level D (N=6) | CLG561, Level E (N=6) | Pretreatment (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arcus lipoides (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 3 | 1 | 3 | 1 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Conjunctivochalasis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 2 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eyelid cyst (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lacrimal disorder (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Optic atrophy (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0
Optic disc disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 3 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Vitreal cells (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitreous degeneration (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 0
Vitreous opacities (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cutis laxa (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.